CLINICAL TRIAL: NCT06519175
Title: Observational Retrospective and Prospective Study of Infantile Lower Limb Malformations and Deformities
Brief Title: Study of Infantile Lower Limb Malformations and Deformities
Acronym: REMEDIA-I
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: Ospedale Pediatrico Bambino Gesù (Unknown); Istituto Giannina Gaslini (Other); Galeazzi Orthopedic Institute (Unknown); Istituto Nazionale Tumori Regina Elena (Unknown); Policlinico San Matteo (Unknown); Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: REMEDIA-I
Record Dates: First submitted 2024-05-06; First posted 2024-07-25 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Deformity of Limb
Keywords: Pediatric orthopedics; Deformity; Patient Reported Outcomes
MeSH Terms: conditions — Congenital Abnormalities | interventions — Conservative Treatment; Single Person; Amputation, Surgical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children and adolescent with lower limb deformities
  Interventions: Other: Conservative treatment; Procedure: Single or multi-stage surgery; Procedure: Amputation

INTERVENTIONS:
Other: Conservative treatment — Patients are provided with physiotherapy support and the provision of prostheses with the goal of ensuring as much walking functionality as possible.
Procedure: Single or multi-stage surgery — Correction of the deformity is pursued by one or more surgical procedures with the timing and the techniques (growth modulation, acute correction, gradual correction, soft tissues procedures, combined techniques) chosen according to the surgeon's preference to achieve the maximum possible walking functionality without orthopedic aids.
Procedure: Amputation — Limb surgery, whether or not associated with realignment or soft-tissue surgery, is performed, aimed at providing the maximum possible walking function through a prosthesis.

SUMMARY:
The skeletal defects of the lower limbs in pediatric age encompass various congenital and acquired conditions that alter bone structure. These alterations can be symmetrical or asymmetrical, with potential consequences such as deformities, short stature, and disability. These condictions may impact not only on the physical and the mental function of the children, but also on their family context.

Management often requires a multidisciplinary approach for early diagnosis and treatment. Deformities are heterogeneous and necessitate a personalized therapeutic plan.

Currently, in pediatric orthopedic surgery there is a lack of an instrument capable of evaluating all these aspects.

The advancement of computer-assisted surgery and artificial intelligence could improve treatment customization and involve patients and families in therapeutic decision-making to prevent complications. This study aims to provide support for clinical practice to promote a systematic, comprehensive, and sequential evaluation of lower limb deformities in developmental age, from which epidemiological data and evidence on treatment approaches used in major referral centers can be extrapolated.

ELIGIBILITY:
Inclusion Criteria:

* Age < 18 years at the time of initial orthopedic evaluation
* Diagnosis of congenital or acquired musculoskeletal deformity to one or both lower limbs
* Presence of informed consent to participate in the study

Exclusion Criteria:

* Refuse to participate in the study by the patient or parent/legal guardian
* Patients with mild paramorphisms not associated with functional limitations

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with congenital or acquired deformity of one or both lower limb diagnosed before skeletal maturity.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Pediatric Outcomes Data Collection Instrument | At baseline (day 0)
  The scores, reported by the child and the caregiver, on the items of the questionnaire, which includes upper extremity (UE), transfer/basic mobility (TBM), happiness (Hap), sports/physical function (SPF), pain/comfort (PC)
Pediatric Outcomes Data Collection Instrument | After 1 year
  The scores, reported by the child and the caregiver, on the items of the questionnaire, which includes upper extremity (UE), transfer/basic mobility (TBM), happiness (Hap), sports/physical function (SPF), pain/comfort (PC)
Clinical examination with complete assessment of lower limbs | At baseline (day 0)
  Full assessment of parameters about lower limb alignment
Clinical examination with complete assessment of lower limbs | After 1 year
  Full assessment of parameters about lower limb alignment
Mental Health | At baseline (day 0)
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health.
Mental Health | After 1 year
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health.

CONTACTS AND LOCATIONS:
Overall Officials: Pierfrancesco Costici, MD, Principal Investigator — Ospedale Pediatrico Bambin Gesù; Giorgio Marrè Brunenghi, MD, Principal Investigator — Istituto Giannina Gaslini; Fabio Verdoni, MD, Principal Investigator — Galeazzi Orthopedic Institute; Roberto Biagini, MD, Principal Investigator — Istituto Nazionale Tumori Regina Elena; Gianluigi Pasta, MD, Principal Investigator — Policlinico San Matteo; Tommaso Bonanzinga, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (7):
- Italy (7):
  - IRCCS Istituto Ortopedico Rizzoli, Bologna
  - Istituto Giannina Gaslini, Genova
  - Galeazzi Orthopedic Institute, Milan
  - Policlinico San Matteo, Pavia
  - Istituto Nazionale Tumori Regina Elena, Roma
  - Ospedale Pediatrico Bambino Gesù, Roma
  - Istituto Clinico Humanitas, Rozzano

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Herring J, Tachdjian's Pediatric Orthopaedics: From the Texas Scottish Rite Hospital for Children, 6th edition. Elsevier, 2020.
- [Background] Sabharwal S. Pediatric Lower Limb Deformities: Principles and Techniques of Management. Springer 2015.
- [Background] Gupta P, Gupta V, Patil B, Verma V. Angular deformities of lower limb in children: Correction for whom, when and how? J Clin Orthop Trauma. 2020 Mar-Apr;11(2):196-201. doi: 10.1016/j.jcot.2020.01.008. Epub 2020 Jan 27. PMID 32099279
- [Background] Chhina H, Klassen AF, Kopec JA, Oliffe J, Iobst C, Dahan-Oliel N, Aggarwal A, Nunn T, Cooper AP. What matters to children with lower limb deformities: an international qualitative study guiding the development of a new patient-reported outcome measure. J Patient Rep Outcomes. 2021 Apr 1;5(1):30. doi: 10.1186/s41687-021-00299-w. PMID 33792793
- [Background] Iobst C. Limb lengthening combined with deformity correction in children with the Taylor Spatial Frame. J Pediatr Orthop B. 2010 Nov;19(6):529-34. doi: 10.1097/BPB.0b013e32833dec43. PMID 20739904
- [Background] Frizziero L, Santi GM, Liverani A, Napolitano F, Papaleo P, Maredi E, Gennaro GLD, Zarantonello P, Stallone S, Stilli S, et al. Computer-Aided Surgical Simulation for Correcting Complex Limb Deformities in Children. Applied Sciences. 2020; 10(15):5181.
- [Background] Blobel B, Ruotsalainen P, Oemig F, Giacomini M, Sottile PA, Endsleff F. Principles and Standards for Designing and Managing Integrable and Interoperable Transformed Health Ecosystems. J Pers Med. 2023 Nov 4;13(11):1579. doi: 10.3390/jpm13111579. PMID 38003894
- [Background] Stuberg W, Temme J, Kaplan P, Clarke A, Fuchs R. Measurement of tibial torsion and thigh-foot angle using goniometry and computed tomography. Clin Orthop Relat Res. 1991 Nov;(272):208-12. PMID 1934735
- [Background] Beighton P, Horan F. Orthopaedic aspects of the Ehlers-Danlos syndrome. J Bone Joint Surg Br. 1969 Aug;51(3):444-53. No abstract available. PMID 5820785
- [Background] Dodwell ER, Pathy R, Widmann RF, Green DW, Scher DM, Blanco JS, Doyle SM, Daluiski A, Sink EL. Reliability of the Modified Clavien-Dindo-Sink Complication Classification System in Pediatric Orthopaedic Surgery. JB JS Open Access. 2018 Oct 23;3(4):e0020. doi: 10.2106/JBJS.OA.18.00020. eCollection 2018 Dec 20. PMID 30882054
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660